CLINICAL TRIAL: NCT03267693
Title: Gastrointestinal Complications in Association With Oropharyngeal and Respiratory Infections in Mechanical Ventilation
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Menna Allah Gamal, Principal Investigator, Assiut University
Other Study IDs: Gastrointestinal tract and VAP
Record Dates: First submitted 2017-08-27; First posted 2017-08-30 (Actual); Last update posted 2017-08-30 (Actual); Status verified 2017-08

CONDITIONS: Ventilator Associated Pneumonia
MeSH Terms: conditions — Pneumonia, Ventilator-Associated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Gastric and oropharyngeal PH — measurement of gastric and oropharyngeal PH and their relation to respiratory and gastrointestinal complication in mechanically ventilated patients

SUMMARY:
Detection of gastrointestinal complications in mechanically ventilated critically ill patients and its relation to oropharyngeal and respiratory infections in relation to oropharyngeal and gastric PH.

DETAILED DESCRIPTION:
Hospital acquired or nosocomial infections continue to be an important cause of morbidity and mortality. The critically ill patient is at particular risk of developing intensive care unit acquired infection, with the lungs being especially vulnerable. Nosocomial bacterial pneumonia occurring after two days of mechanical ventilation is referred to as ventilator associated pneumonia, and is the most common nosocomial infection seen in the intensive care unit. Intubation of the trachea and mechanical ventilation is associated with a 7-fold to 21-fold increase in the incidence of pneumonia and up to 28% of patients receiving mechanical ventilation will develop this complication. Its development is associated with an attributable increase in morbidity and mortality. Ventilator associated pneumonia (VAP) is defined as nosocomial pneumonia occurring in a patient after 48 hours of mechanical ventilation via a tracheal or tracheostomy tube. It is commonly classified as either early onset (occurring within 96 hours of start of mechanical ventilation) or late onset (.96 hours after start of mechanical ventilation). It is a common condition, difficult to diagnose accurately, and expensive to treat. Its development prolongs a patient's stay in the intensive care unit (ICU), and is associated with significant morbidity and mortality. Most cases seem to result from aspiration of pathogenic material that commonly colonises the oropharyngeal airways of the critically ill. Simple measures to decrease the incidence of aspiration or reduce the burden of colonisation of the oropharynx may aid in the prevention of ventilator associated pneumonia. VAP is the infection that occurs 48 hours after intubation, which was not incubated during the period of the patient's admission, and 72 hours after extubation.

The gastrointestinal tract is believed to play an important role in ventilator-associated pneumonia (VAP), because during critical illness the stomach often is colonized with enteric Gram-negative bacteria. These are the same bacteria that frequently are isolated from the sputum of patients with VAP.

This is known as the "gastropulmonary hypothesis" and it postulates the following sequence. First, the stomach is colonized by potentially pathogenic microorganisms, either from an exogenous source (contaminated liquid injected into a nasogastric tube), or from an endogenous source (Detection of gastrointestinal complications in mechanically ventilated critically ill patients and its relation to oropharyngeal and respiratory infections in relation to oropharyngeal and gastric PH duodenogastric reflux). This is followed by retrograde colonization of the oropharynx . Finally, the lower respiratory tract is colonized from sustained microaspiration of contaminated oropharyngeal (or gastric) secretions around the endotracheal tube cuff.

The Role of Gastric pH on the Incidence of VAP

Under fasting conditions, gastric sterility is maintained by an acidic pH. Clinical evidence suggests that a gastric pH of 3.5 prevents bacterial colonization, whereas a pH 4.0 is associated with clinically important bacterial colonization and a higher incidence of nosocomial pneumonia.

Critically-ill patients with either respiratory failure requiring mechanical ventilation or coagulopathy are at increased risk for clinically important, stress-related GI bleeding .This has been associated with a significantly higher mortality rate, compared to patients without evidence of bleeding (48.5 vs 9.1%, p _ 0.001).

Giving that such patients show an increasing risk of important gastrointestinal (GI) bleeding, stress-ulcer prophylaxis (SUP) has been recommended for the prevention of upper GI hemorrhage. SUP strategy rely on drugs that block the secretion of gastric acid and increase the gastric pH (histamine-2-receptor antagonists - H2RA, and proton pump inhibitor - PPI) and those that does not alter gastric pH (sucralfate). The increase of gastric pH leads to bacterial overgrowth and potential colonization of trachea determining a higher risk of VAP.

ELIGIBILITY:
Inclusion Criteria:

* all critically ill mechanically ventilated patients between 18 and 70 years

Exclusion Criteria:

* patients take drugs affect gastric and oropharyngeal PH such as antacids, proton pump inhibitors, H2 receptor antagonists

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: male and female patients between 18 and 70 years in ICU units on mechanical ventilator
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-09 (Estimated); Primary Completion 2018-09 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
measurement of gastric and oropharyngeal ph in mechanically ventilated patients | 30 minutes
  correlation between gastric and oropharyngeal ph and presence of gastrointestinal and respiratory complications in mechanically ventilated patients

REFERENCES:
- [Background] Hunter JD. Ventilator associated pneumonia. Postgrad Med J. 2006 Mar;82(965):172-8. doi: 10.1136/pgmj.2005.036905. PMID 16517798